CLINICAL TRIAL: NCT07079904
Title: Comparison of Single Operator Laser-assisted Ultrasound-guided Peripheral Vein Cannulation With Traditional Ultrasound Guidance in Patients Receiving Cardiac Surgery
Brief Title: Laser-assisted Ultrasound-guided Peripheral Vein Cannulation in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shuai Wang, Deputy Chief Nurse, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KY20250527-01
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ultrasonography, Interventional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Other): In group T, ultrasound-guided peripheral vein cannulation was performed using dynamic needle tip positioning technique.
  Interventions: Other: Ultrasound Guided Peripheral Vein Catheterization With or Without Laser-Assisted.
- Group L (Experimental): In group L, ultrasound-guided peripheral vein cannulation was performed using dynamic needle tip positioning technique with laser-assisted.
  Interventions: Other: Ultrasound Guided Peripheral Vein Catheterization With or Without Laser-Assisted.

INTERVENTIONS:
Other: Ultrasound Guided Peripheral Vein Catheterization With or Without Laser-Assisted. — In group T, ultrasound-guided peripheral vein cannulation was performed using dynamic needle tip positioning technique. In group L, ultrasound-guided peripheral vein cannulation was performed using dynamic needle tip positioning technique with laser-assisted.

SUMMARY:
The aim of this clinical trial is to investigate the advantages of single-operator laser-assisted ultrasound-guidance comparing with traditional ultrasound guidance in peripheral venous catheterization.The primary question addressed is whether single-operator laser-assisted ultrasound-guidance could improve the first-attempt success rate of peripheral venous catheterization compared with traditional ultrasound guidance.

DETAILED DESCRIPTION:
One hundred patients receiving cardiac surgery were randomized into two groups control group (group T, 50 patients), and experimental group (group L, 50 patients). In group T, ultrasound-guided short-axis out-of-plane technique with dynamic needle tip positioning is employed. The operator holds the puncture needle in the right hand at an angle of approximately 30-40° to the skin, and inserts the needle along the projection path of the laser on the body surface at a distance of about 0.5 cm from the probe. Under direct visualization, the needle tip is inserted into the blood vessel, and then the probe is slowly moved along the course of the vein to keep the needle tip directly above the vessel, thereby obtaining the optimal axial cross-section with this as the axis. After observing the high-echo needle tip displayed in the blood vessel on the ultrasound image, keep the puncture needle still and move the ultrasound probe until it disappears. Slowly advance the puncture needle so that the needle tip is always located in the center of the blood vessel during the puncture process. After observing the needle body reaching the blood vessel, withdraw the needle core, and then insert the catheter into it. In group L, an nurse prepares the equipment as follows before the patient enters the operating room: the mechanical arm is fixed near the operating table, and the laser emitter is attached is attached nearby. The tightness is adjusted to ensure a tighter fit between the probe and its housing. The ultrasound probe is then placed over the middle of the elbow and slightly moved so that the central auxiliary line on the screen passes through the center of the blood vessel. After the image is saved, another nurse measures the diameter and depth of the vein. The first point under the middle of the ultrasound probe is marked with a sterile marker pen. The probe is then moved 1.0 cm proximally, and the second point is marked in the same way. The probe is fixed to the skin at an angle of approximately 75°. After turning on the laser, the laser beam is aligned to pass through the middle mark of the ultrasound probe (centered on the vein lumen) and the two marked points: the laser beam thus becomes the skin projection of the venous anatomical path. At this point, the probe is fixed with the mechanical arm, and the needle is held in the right hand. Finally, the height of the ultrasound screen is adjusted to be level with the operator's eyes to reduce head and neck movement and facilitate guidance. Then, venous catheterization was completed with the "dynamic needle tip positioning" method.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-80 years
2. BMI 18-30 kg/m²
3. ASA classification 1-4

Exclusion Criteria:

1. infection or hematoma at the puncture site
2. patients mentally unstable or unable to cooperate
3. patient refused to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
First-attempt success rate | immediately after the intervention
  The completion of the cannulation was defined as the presentation of the arterial waveform on the monitor.

SECONDARY OUTCOMES:
The overall rate of successful catheterizations The overall rate of successful catheterizations | immediately after the intervention
  Counted at the completion of the procedure and calculated during the data collation phase
The number of unintentional penetration of the posterior wall of the venous | From the beginning of puncture to completion of catheterization
  Counted during the procedure and calculated during the data collation phase
The procedure time to success within the first attempt | From the beginning of puncture to completion of catheterization in the first attempt
  Counted during the procedure
Overall procedure time | immediately after the procedure
  Counted during the procedure and calculated during the data collation phase
The average number of adjustments | From the beginning of puncture to completion of catheterization
  Counted during the procedure and calculated during the data collation phase
The midmost rate of first attempt | After the first needle insertion
  Ultrasound images were stored and evaluated after the whole procedure.
The first needle-tip position | After the first needle insertion
  Ultrasonic images were stored and evaluated by quadrant method after the whole procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Wang, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No